CLINICAL TRIAL: NCT02422667
Title: iCORE: Collaborative Orthopedics Outcomes Registry
Acronym: iCORE
Status: Withdrawn | Type: Observational
Why Stopped: Study cancelled - no results
Sponsor: SCRI Development Innovations, LLC (Other)
Responsible Party: Sponsor
Other Study IDs: SCRI HEOR_03
Record Dates: First submitted 2015-04-14; First posted 2015-04-21 (Estimated); Last update posted 2023-12-05 (Actual); Status verified 2020-08

CONDITIONS: Arthroplasty, Replacement, Hip; Arthroplasty, Replacement, Knee
Keywords: Orthopedics; Outcome Assessment

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Patient Registry — Orthopedic Data Registry

SUMMARY:
The goal of this registry is to review the data collected and research ways to improve patient safety, quality of care, and medical decision-making, reduce medical spending, and help advance orthopedic science and bioengineering.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Patients requested to be seen by an orthopedic surgeon participating in the iCORE Registry.
* Patient must have the ability to understand the nature of the registry and give written informed consent.

Exclusion Criteria:

* There are no exclusion criteria for this Outcomes Registry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients 18 years and older who undergo hip and/or knee arthroplasty. Patient must have the ability to understand the nature of the registry and give written informed consent.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Quality Improvement | 10 years
Treatment Patterns | 5 years
Healthcare Utilization | 5 years

SECONDARY OUTCOMES:
Humanistic Outcomes | 10 years
Economic Outcomes | 10 years

CONTACTS AND LOCATIONS:
Overall Officials: David K DeBoer, MD, Principal Investigator — SJRI/SCRI
Locations (1):
- SCRI, Nashville, Tennessee, United States